CLINICAL TRIAL: NCT04274829
Title: Predictive Factors of Lymph Node Metastasis in Patients With Papillary Microcarcinoma of the Thyroid
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Assistant Professor, University of Cagliari
Other Study IDs: MICRO-PTC-LN
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Thyroid Cancer; Lymph Node Metastases
MeSH Terms: conditions — Thyroid Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PTMC: Patients with papillary microcarcinoma of the thyroid
  Interventions: Procedure: Thyroidecomt and lymphectomy

INTERVENTIONS:
Procedure: Thyroidecomt and lymphectomy — Patients underwent total thyroidectomy or lobectomy associated to lymph node sampling or neck lymphectomy

SUMMARY:
Papillary thyroid microcarcinoma (PTMC), defined as a tumor with larger diameter ≤ 1 cm, is considered a tumor with an indolent course and an excellent prognosis. Nevertheless, the incidence of lymph node metastasis in PTMC is not negligible, reaching up to 65% in some series. The aim of this study was to assess the incidence of lymph node metastasis in patients with PTMC and to evaluate predictive factors for lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

Patients with papillary microcarcinoma of the thyroid

Exclusion Criteria:

Patients with thyroid nodules > 1 cm; incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with papillary thyroid carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Incidence of lymph node metastasis | 1 year
  To define the incidence of lymph node metastasis in patients with papillary microcarcinoma

SECONDARY OUTCOMES:
Predicrive factors of lymph node metastasis | 1 year
  To assesss predictive factors of lymph node metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Cagliari, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Medas F, Canu GL, Cappellacci F, Boi F, Lai ML, Erdas E, Calo PG. Predictive Factors of Lymph Node Metastasis in Patients With Papillary Microcarcinoma of the Thyroid: Retrospective Analysis on 293 Cases. Front Endocrinol (Lausanne). 2020 Aug 25;11:551. doi: 10.3389/fendo.2020.00551. eCollection 2020. PMID 32982963